CLINICAL TRIAL: NCT01111747
Title: Regeneration of the Patellar Tendon After Harvesting Its Central Third With Platelet-rich Plasma. Prospective and Randomized Study.
Brief Title: Patellar Tendon Regeneration With Platelet-rich Plasma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Instituto de Ortopedia e Traumatologia - HCFMUSP - São Paulo, Brazil (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0162/08; CaPPesqHCFMUSP 0162/2008 (Other: São Paulo University)
Record Dates: First submitted 2010-04-26; First posted 2010-04-28 (Estimated); Last update posted 2012-03-14 (Estimated); Status verified 2010-04

CONDITIONS: Knee Instability
Keywords: platelet-rich plasma; patellar ligament; regeneration; growth substances
MeSH Terms: interventions — Intercellular Signaling Peptides and Proteins; Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRP (Experimental): In this group PRP will be used in the patellar tendon donor site.
  Interventions: Procedure: Platelet-rich plasma
- Control (Sham Comparator): In this group PRP will not be aded to the patellar tendon donor site
  Interventions: Procedure: Control group

INTERVENTIONS:
Procedure: Platelet-rich plasma — Intra-operative use of platelet-rich plasma in the patellar tendon after harvesting its central third for ACL reconstruction.
  Other Names: PRP; platelet gel; platelet concentrate; growth factors concentrate; plasma rich in growth factors
  Arms: PRP
Procedure: Control group — In this group PRP will not be added to the patellar tendon donor site at the end of ACL reconstruction.
  Other Names: PRP; platelet-rich plasma; platelet gel; platelet concentrate; growth factors concentrate; plasma rich in growth factors
  Arms: Control

SUMMARY:
The central third of the patellar tendon is used as a donor site for anterior cruciate ligament (ACL) reconstruction. After months or years the harvest site partially regenerates. The regeneration process is accomplished by biological mechanisms,including cells and proteins known as growth factors. The platelets are natural reservoirs of growth factors, and a platelet concentrate known as Platelet-Rich Plasma (PRP) has a three to five fold increase in growth factors. The hypothesis of the study is that the PRP can improve the regeneration of the patellar tendon.

The platelets are obtained from the patient's blood through a filtration system called apheresis, with the use of 250 milliliters of blood, with a sterile system. All the others components of blood (red cells, plasma, white cells) returns to the patient. The PRP is then applied in the harvest site on the patellar tendon, at the end of ACL reconstruction.

The patients are randomized in two groups, one with the use of PRP and the other group without PRP. This information for the patients will be granted just at the end of the research. After the surgery the rehabilitation protocol is the same for both groups. An isokinetic testing is done before the surgery and after six months. Questionnaires about the knee function are asked before the surgery and after six months. A magnetic resonance imaging is performed after six months to evaluate the tendon regeneration.

ELIGIBILITY:
Inclusion Criteria:

* indication of anterior cruciate ligament surgery with patellar ligament
* skeletal maturity

Exclusion Criteria:

* other knee ligament injuries
* severe chondral lesions
* osteoarthritis
* non-compliance to the rehabilitation
* previous surgery in the affected knee
* reoperation during the time of the study for an unrelated condition
* infection

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 27 (Actual)
Dates: Start 2008-11; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the patellar tendon regeneration with magnetic resonance imaging. | Six months
  Six months after the surgery a magnetic resonance imaging will be done to evaluate the regeneration of the patellar tendon donor site. The area of the gap, related to the tendon harvest, will be measured and compared between the groups.

SECONDARY OUTCOMES:
Isokinetic testing and questionaires. | Six months
  Six months after the surgery, patients will answer to questionaires about their knee function and do an isokinetic testing to evaluate their muscle strength. The results will be compared between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Adriano M Almeida, MD, Principal Investigator — Instituto de Ortopedia e Traumatologia - HCFMUSP - São Paulo, Brazil; Arnaldo J Hernandez, MD, PhD, Study Director — Instituto de Ortopedia e Traumatologia - HCFMUSP - São Paulo, Brazil

REFERENCES:
- [Background] Kartus J, Movin T, Papadogiannakis N, Christensen LR, Lindahl S, Karlsson J. A radiographic and histologic evaluation of the patellar tendon after harvesting its central third. Am J Sports Med. 2000 Mar-Apr;28(2):218-26. doi: 10.1177/03635465000280021301. PMID 10750999
- [Background] Meisterling RC, Wadsworth T, Ardill R, Griffiths H, Lane-Larsen CL. Morphologic changes in the human patellar tendon after bone-tendon-bone anterior cruciate ligament reconstruction. Clin Orthop Relat Res. 1993 Apr;(289):208-12. PMID 8472418
- [Background] Svensson M, Kartus J, Ejerhed L, Lindahl S, Karlsson J. Does the patellar tendon normalize after harvesting its central third?: a prospective long-term MRI study. Am J Sports Med. 2004 Jan-Feb;32(1):34-8. doi: 10.1177/0363546503258935. PMID 14754721
- [Background] Anaguchi Y, Yasuda K, Majima T, Tohyama H, Minami A, Hayashi K. The effect of transforming growth factor-beta on mechanical properties of the fibrous tissue regenerated in the patellar tendon after resecting the central portion. Clin Biomech (Bristol). 2005 Nov;20(9):959-65. doi: 10.1016/j.clinbiomech.2005.05.012. PMID 16055249
- [Background] Anitua E, Andia I, Ardanza B, Nurden P, Nurden AT. Autologous platelets as a source of proteins for healing and tissue regeneration. Thromb Haemost. 2004 Jan;91(1):4-15. doi: 10.1160/TH03-07-0440. PMID 14691563
- [Background] Spindler KP, Nanney LB, Davidson JM. Proliferative responses to platelet-derived growth factor in young and old rat patellar tendon. Connect Tissue Res. 1995;31(2):171-7. doi: 10.3109/03008209509028405. PMID 15612333
- [Background] Molloy T, Wang Y, Murrell G. The roles of growth factors in tendon and ligament healing. Sports Med. 2003;33(5):381-94. doi: 10.2165/00007256-200333050-00004. PMID 12696985
- [Background] Aspenberg P. Stimulation of tendon repair: mechanical loading, GDFs and platelets. A mini-review. Int Orthop. 2007 Dec;31(6):783-9. doi: 10.1007/s00264-007-0398-6. Epub 2007 Jun 22. PMID 17583812
- [Background] Rodeo SA, Potter HG, Kawamura S, Turner AS, Kim HJ, Atkinson BL. Biologic augmentation of rotator cuff tendon-healing with use of a mixture of osteoinductive growth factors. J Bone Joint Surg Am. 2007 Nov;89(11):2485-97. doi: 10.2106/JBJS.C.01627. PMID 17974893
- [Background] Sanchez M, Anitua E, Azofra J, Andia I, Padilla S, Mujika I. Comparison of surgically repaired Achilles tendon tears using platelet-rich fibrin matrices. Am J Sports Med. 2007 Feb;35(2):245-51. doi: 10.1177/0363546506294078. Epub 2006 Nov 12. PMID 17099241